CLINICAL TRIAL: NCT00226707
Title: A 6-Week Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel Group Study to Investigate the Efficacy and Safety of Pimecrolimus Cream 1% in Patients With Mild-to-Moderate Chronic Hand Dermatitis Followed by a 6-Week Open-Label Phase to Assess the Safety of Pimecrolimus Cream 1%
Brief Title: Pimecrolimus Cream 1% in Patients (18 Years of Age and Over) With Mild to Moderate Chronic Hand Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981M2301
Record Dates: First submitted 2005-09-26; First posted 2005-09-27 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Chronic Hand Dermatitis
Keywords: Chronic hand dermatitis, pimecrolimus, dermatitis
MeSH Terms: conditions — Dermatitis | interventions — pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus Cream 1%
  Other Names: Elidel

SUMMARY:
Topical steroids are standard of care for Chronic Hand Dermatitis, but long-term use is associated with adverse effects. This study will assess the efficacy and safety of pimecrolimus cream 1% in patients with mild-to-moderate chronic hand dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who are outpatients at baseline (Day 1)
* Patients must be 18 years of age or above
* Patients must have chronic hand dermatitis based upon clinical diagnosis with mild to moderate dermatitis of the target hand at baseline, as defined by an Investigator's Global Assessment score of 2 (mild) or 3 (moderate).
* Patients must have been informed of the study procedures and medication and have given their written informed consent

Exclusion Criteria:

* - Women who are pregnant or who are breast-feeding.
* Patients who have received systemic corticosteroids (i.e., oral, intravenous, intra-articular, rectal, intramuscular) within one month prior to first application of study medication.
* Patients who have received phototherapy (e.g., UVB, PUVA) or systemic therapy (e.g., immunosuppressants, cytostatics) known or suspected to have an effect on hand dermatitis within at least one month prior to first application of study medication.
* Patients who have received pimecrolimus cream 1% or tacrolimus ointment 0.1% or 0.03% within 14 days prior to first application of study medication.
* Patients who were treated with topical therapy (e.g., tar, topical corticosteroids, Burrows solution soaks) known or suspected to have an effect on hand dermatitis within 7 days prior to first application of trial medication.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 652
Dates: Start 2004-07; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Investigators Global Assessment (IGA) of the target hand at day 43 or at time of early discontinuation.

SECONDARY OUTCOMES:
IGA of the non-target hand
Itching/burning assessment for the target and non-target hand
Non-key signs of hand dermatitis (vesiculation, oozing/crusts, edema/population, lichenification) at each study visit
Work productivity and activity impairment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Study Chair — Novartis Pharmaceuticals